CLINICAL TRIAL: NCT05460585
Title: Comparison of Cerebral Oxygenation Values in Healthy Adults
Brief Title: Cerebral Oxygenation Values in Healthy Adults Volunteers Measured With RheoPatch and NIRO-200NX
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-D0083
Record Dates: First submitted 2022-07-05; First posted 2022-07-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy; Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Cerebral oximetry using Rheopatch — On the study visit, baseline demographic data (age and gender, BMI) are collected. In supine position the sensor patches (left and right) of the device are applied to the forehead and the cerebral oxymetry values are recorded during 120sec. The sensor patches are then removed and the patches of the second device are applied on the same position on the forehead and the measurement is carried out as described before. For the first measurement of each sensor, a total of 5 minutes equilibration and sensor output power adjustment is allowed. A total of 10 measurements are taken, 5 with each device.
  The volunteer is then placed in Trendelenburg position and another 4 measurements are made (2 with each device) as previously described.
Device: Cerebral oximetry using NIRO-200NX — On the study visit, baseline demographic data (age and gender, BMI) are collected. In supine position the sensor patches (left and right) of the device are applied to the forehead and the cerebral oxymetry values are recorded during 120sec. The sensor patches are then removed and the patches of the second device are applied on the same position on the forehead and the measurement is carried out as described before. For the first measurement of each sensor, a total of 5 minutes equilibration and sensor output power adjustment is allowed. A total of 10 measurements are taken, 5 with each device.
  The volunteer is then placed in Trendelenburg position and another 4 measurements are made (2 with each device) as previously described.

SUMMARY:
Noninvasive measurement of cerebral tissue oxygen saturation levels by near infrared spectroscopy (NIRS) is clinical routine in perioperative medicine. One of the main technical challenges of NIRS measurements is to eliminate the influence of signals of the skin and skull. A new device (RheoPatch, Luciole Medical AG, Zurich) has been developed by a company that also developed an intracranial NIRS probe, which allowed measurements directly in the brain and thus improved algorithms for elimination of the extracranial signals. The investigators aim to determine baseline values and performance of the new device (RheoPatch) compared with a more established NIRS device (NIRO-200NX, Hamamatsu Phototonics, Hamamatsu City, Japan)

DETAILED DESCRIPTION:
Primary objective is to compare the RheoPatch NIRS device with the NIRO-200NX NIRS device in volunteers at rest in supine position. As secondary objectives, repeatability of the measurements will be tested with optode reapplications. With measurements in Trendelenburg position, the investigators evaluate the influence of body (head) position on the NIRS signals.

Primary outcome are the baseline values of cerebral oxygenation levels measured by RheoPatch (SbtO2 (%)) and NIRO-200NX (Tissue oxygenation index: TOI (%)).

Secondary endpoints are the repeatability of the measurements with sensor reapplications (coefficient of repeatability, 5 repeats with each device) and changes of the measurements of cerebral oxygenation saturation level in the Trendelenburg position.

Measurements of baseline cerebral oxygenation values are obtained in supine position with 10 measurements, alternating between devices. Combined with 5 min measurement phase for equilibration and power adjustment, this will require 33 minutes per participant.

ELIGIBILITY:
Inclusion Criteria:

Subjects fulfilling all of the following inclusion criteria are eligible for the investigation:

* Informed Consent signed by the subject
* Subjective good health

Exclusion Criteria:

The presence of any one of the following exclusion criteria will lead to the exclusion of the subject

* Age (<18, > 65 yrs.)
* Forehead skin disease
* Allergy to skin contacting components of NIRS-sensors
* Known cerebrovascular and heart diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The project population consists of volunteers in subjective good health. Volunteers are chosen to minimize the effect of diseases on the measurements, as the investigators are interested in baseline measurement values and repeatability.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen saturation level | One day
  Primary endpoint is the cerebral oxygen saturation level measured by RheoPatch (SbtO2 (%)) and NIRO-200NX (Tissue oxygenation index: TOI (%)). This is the value used for clinical decision making in the daily routine when NIRS measurement devices are used in perioperative medicine or intensive care applications and therefore the most relevant value.

SECONDARY OUTCOMES:
Changes of the measurements of cerebral oxygenation saturation level (SbtO2 (%) and TOI (%)) | One day
  SbtO2 and TOI changes are measured
nTHI_NIRO | One day
  Normalized tissue hemoglobin index: nTHI (absolute value in arbitrary unit)
ΔO2Hb_NIRO | One day
  Oxygenated hemoglobin change: ΔO2Hb (μmol/L)
ΔHHb_NIRO | One day
  Deoxygenated hemoglobin change: ΔHHb (μmol/L)
ΔcHb_NIRO | One day
  Total hemoglobin change: ΔcHb (μmol/L)
aH2O_RP | One day
  Absolute concentration of brain tissue water: aH2O (mmol/L)
aHbDeoxy_RP | One day
  Absolute concentration of deoxygenated hemoglobin: aHbDeoxy (μmol/L)
aHbOxy_RP | One day
  Absolute concentration of oxygenated hemoglobin: aHbOxy (μmol/L)
aHbTotal_RP | One day
  Absolute concentration of total hemoglobin: aHbTotal (μmol/L)
ΔO2Hb_RP | One day
  Oxygenated hemoglobin change: ΔO2Hb (μmol/L)
ΔHHb_RP | One day
  Deoxygenated hemoglobin change: ΔHHb (μmol/L)
ΔcHb_RP | One day
  Total hemoglobin change: ΔcHb (μmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Erdoes, MD PhD, Study Chair — University of Bern
Locations (1):
- Dep. Anesthesiology and Pain Therapy, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No